CLINICAL TRIAL: NCT00222066
Title: Comparison Between Abstention and Intrauterine Aspiration in the Treatment of Anechoic Fetal Ovarian Cysts to Prevent Ovarian Torsion
Brief Title: Effect of Fetal Ovarian Cyst Aspiration to Prevent Torsion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Pr Franck Perrotin, CHRU de Tours
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OV-UTERO 2000
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2006-09

CONDITIONS: Ovarian Cyst; Ultrasonography Prenatal
Keywords: Aspiration; Fetal ovarian cyst; Ovarian torsion
MeSH Terms: conditions — Ovarian Cysts; Neonatal ovarian cyst; Ovarian Torsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Fetal ovarian cyst aspiration performed as soon as possible
  Interventions: Procedure: Fetal ovarian cyst aspiration
- 2 (No Intervention): Expectative

INTERVENTIONS:
Procedure: Fetal ovarian cyst aspiration — Fetal ovarian cyst aspiration performed under ultrasound guidance and maternal local anesthesia
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether prenatal ovarian cyst aspiration is effective and safe to prevent perinatal ovarian torsion.

DETAILED DESCRIPTION:
With the widespread use of routine sonography during pregnancy, the incidence of fetal ovarian cysts detected in utero has increased in the past decades. However

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women having an uneventful single pregnancy and a female fetus diagnosed with anechoic ovarian cyst (diameter at least 30mm)

Exclusion Criteria:

* Multiple pregnancy
* Complicated pregnancy (PE, diabetes, PROM, fetal malformation)
* Echoic cyst (fluid debris level, septated, retracting clot, globally echoic)
* Unability to give informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2001-06; Primary Completion 2007-01 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To avoid neonatal surgery | 3 months after birth

SECONDARY OUTCOMES:
Ultrasound pattern of neonatal ovarian cyst | 3 months after birth
Maternal and fetal/neonatal safety of prenatal ovarian cyst aspiration | 3 months after birth

CONTACTS AND LOCATIONS:
Overall Officials: Franck Perrotin, MD--PhD, Principal Investigator — Tours University Hospital
Locations (3):
- France (3):
  - Olympe de Gouges Women Health Centre, Bretonneau University Hospital, Tours, Centre-Val de Loire
  - CHU de Nantes, Nantes, Loire Atl
  - CHU de Caen, Caen

REFERENCES:
- [Background] Perrotin F, Potin J, Haddad G, Sembely-Taveau C, Lansac J, Body G. Fetal ovarian cysts: a report of three cases managed by intrauterine aspiration. Ultrasound Obstet Gynecol. 2000 Dec;16(7):655-9. doi: 10.1046/j.1469-0705.2000.00247.x. PMID 11169374
- [Background] Perrotin F, Roy F, Potin J, Lardy H, Lansac J, Body G. [Ultrasonographic diagnosis and prenatal management of fetal ovarian cysts]. J Gynecol Obstet Biol Reprod (Paris). 2000 Apr;29(2):161-9. French. PMID 10790628